CLINICAL TRIAL: NCT00416429
Title: Medroxyprogesterone, Interferon Alpha-2a, Interleukin 2 or Combination of Both Cytokines in Patients With Metastatic Renal Carcinoma of Intermediate Prognosis [PERCY QUATTRO]
Brief Title: Medroxyprogesterone or Interferon and/or Aldesleukin in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000468571; LEONB-PERCY-QUATTRO; EU-20605; LEONB-ET99-058; ROCHE-LEONB-PERCY-QUATTRO; CHIRON-LEONB-PERCY-QUATTRO
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon alpha-2; Medroxyprogesterone

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alpha-2a
Drug: medroxyprogesterone

SUMMARY:
RATIONALE: Medroxyprogesterone may help shrink or slow the growth of kidney cancer. Interferon may interfere with the growth of tumor cells. Aldesleukin may stimulate white blood cells to kill tumor cells. It is not yet known whether giving medroxyprogesterone, interferon, or aldesleukin alone is more effective than giving interferon together with aldesleukin in treating kidney cancer.

PURPOSE: This randomized phase III trial is studying medroxyprogesterone, interferon, or aldesleukin to see how well they work when given alone compared to interferon combined with aldesleukin in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall survival of patients with metastatic renal cell adenocarcinoma treated with medroxyprogesterone vs recombinant interferon alfa-2a and/or aldesleukin.

Secondary

* Determine the objective response rate (complete and partial) of patients treated with these regimens.
* Determine the progression-free survival of patients treated with these regimens.
* Determine the toxicity of these regimens in these patients.
* Evaluate the quality of life of patients before and after induction treatment with these regimens (week 10).

OUTLINE: This is a randomized, controlled, open-label, multicenter study. Patients are randomized to 1 of 4 treatment arms.

* Arm I (medroxyprogesterone): Patients receive oral medroxyprogesterone once daily for 12 weeks. Patients may receive a second 12-week course in the presence of responding or stable disease. Quality of life is assessed at baseline and at weeks 12 and 24.
* Arm II (recombinant interferon alfa-2a): Patients receive recombinant interferon alfa-2a subcutaneously (SC) 3 times weekly for 12 weeks. Patients may receive a second 12-week course in the presence of responding or stable disease. Quality of life is assessed as in arm I.
* Arm III (aldesleukin): Patients receive aldesleukin SC twice daily on days 1-5, 8, 9, 15, 16, 22, and 23 and once daily on days 10-12, 17-19, and 24-26. Courses repeat beginning in weeks 6, 13, and 20. Quality of life is assessed at baseline and at weeks 10 and 24.
* Arm IV (recombinant interferon alfa-2a and aldesleukin): Patients receive recombinant interferon alfa-2a as in arm II and receive aldesleukin as in arm III. Quality of life is assessed as in arm III.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 456 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell adenocarcinoma, meeting 1 of the following criteria:

  * More than 1 metastatic site and good performance status (Karnofsky score 80-100%)
  * Sole metastatic site with Karnofsky score = 80%

    * Karnofsky 90% or 100% not eligible
  * No combination of several metastatic sites and liver metastases and a time interval from primary tumor to metastases of < 1 year
* Nonmeasurable disease and/or few numbers of lesions must be confirmed histologically and as progressive disease
* The following metastases are allowed:

  * Lung with or without mediastinum lymph nodes
  * Bone
  * Pleura (solid or liquid with positive cytology)
  * Thoracic lymph nodes
  * Abdominal lymph nodes
  * Superficial lymph nodes
  * Liver
  * Subcutaneous skin/tissue
  * Contralateral kidney
  * Nephrectomy site
  * Other organs
* Prior metastases allowed provided the following criteria are met:

  * Evidence of progressive disease within the past 3 months
  * Metastases evaluated by noninvasive methods
* No evidence of active brain metastases

  * Prior brain metastases allowed provided all of the following criteria are met:

    * Disease is stable
    * Reductive therapy (surgery or radiotherapy) completed at least 3 weeks prior to study entry
    * Metastases have not progressed (confirmed by CT scan or MRI)
    * No concurrent corticosteroids required

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Creatinine < 1.8 mg/dL
* Hematocrit ≥ 30%
* WBC ≥ 4,000/mm^3
* Platelet count ≥ 120,000/mm^3
* Bilirubin normal
* LVEF ≥ 50%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HIV positivity
* No severe infection requiring antibiotic therapy
* No chronic hepatitis
* No severe lung, liver or kidney condition that would preclude study treatment
* No hepatitis B surface antigen positivity
* No severe neuropsychiatric condition or epilepsy
* No serious thromboembolitic disorder
* No severe cardiac dysfunction (e.g., congestive heart failure, uncontrolled hypertension, serious arrhythmia, or coronary disease)
* No other prior or concurrent primary malignancies except for basal cell skin cancer or carcinoma in situ of the cervix
* No geographical, psychological, or familial condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* More than 6 weeks since prior wide-field radiotherapy
* No prior systemic chemotherapy
* No prior organ transplantation
* No prior cytokines
* No concurrent hormonal therapy
* No concurrent anticancer chemotherapy
* No concurrent corticosteroids
* No other concurrent immunotherapy
* No other concurrent investigational agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Objective response rate (complete and partial)
Progression-free survival
Toxicity
Quality of life in week 10

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Negrier, MD, Study Chair — Centre Leon Berard

REFERENCES:
- [Result] Negrier S, Perol D, Ravaud A, Chevreau C, Bay JO, Delva R, Sevin E, Caty A, Escudier B; French Immunotherapy Intergroup. Medroxyprogesterone, interferon alfa-2a, interleukin 2, or combination of both cytokines in patients with metastatic renal carcinoma of intermediate prognosis: results of a randomized controlled trial. Cancer. 2007 Dec 1;110(11):2468-77. doi: 10.1002/cncr.23056. PMID 17932908